CLINICAL TRIAL: NCT07294404
Title: Effectiveness of Orthokeratology and Peripheral Retinal Refraction Changes
Brief Title: Peripheral Relative Refractive Power of Orthokeratology Lenses
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OK RPR
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: orthokeratology — All participants will be fitted with orthokeratology lenses of the same design. The primary objective is to assess changes in relative peripheral retinal refraction before and after lens wear.

SUMMARY:
Orthokeratology (OK) has been demonstrated to be an effective intervention for slowing axial elongation in children with myopia. The proposed mechanism of action is the induction of peripheral myopic defocus, which reduces relative peripheral hyperopia on the retina.

This study aims to evaluate changes in relative peripheral retinal refraction before and after OK lens wear using wide-field multispectral retinal refractive topography. The study will also investigate the relationship between these retinal refractive changes and the effectiveness of OK in controlling axial elongation.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 15 years old
* myopia of -4.00D or lower,
* regular astigmatism ≤1.50D and non-regular astigmatism ≤1.00D
* intraocular pressure ≤21mmHg
* understand the purpose of the study and have good hygiene and regular follow-up

Exclusion Criteria:

* unilateral
* immunocompromised subjects with systemic diseases (such as acute or chronic sinusitis, diabetes mellitus, Down syndrome, rheumatoid arthritis, psychiatric patients, etc.)
* complicated with other eye diseases that affect OK lens wearing, such as dacryocystitis, blepharitis and other inflammation, glaucoma, etc.
* BCVA more than 1.0
* children with corneal curvature less than 40.00D or higher than 46.00D.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 8 to 15 years with myopia who are eligible for and fitted with orthokeratology lenses. Participants must demonstrate the ability to maintain adequate compliance with lens wear and follow-up requirements.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Changes in axial length growth(ALG) | Change from baseline in axial length at 12 months
  Axial length will be measured using an ocular biometer (AL-Scan, NIDEK, Japan). Axial length growth (ALG) will be defined as the difference between the 1-year measurement and baseline.

SECONDARY OUTCOMES:
Change in Relative Peripheral Retinal Refraction | Baseline (pre-lens wear), 1 month, 6 months, and 12 months after orthokeratology lens wear.
  Retinal refractive power will be measured using multispectral retinal refractive topography. Relative peripheral retinal refraction will be calculated as the difference between peripheral and central retinal refractive power. Changes from pre- to post-orthokeratology lens wear will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaoyan Yang, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No